CLINICAL TRIAL: NCT00414206
Title: A Phase II Randomized, Double-Masked, Study Comparing the Safety and Efficacy of ATG003 in Patients With Neovascular ("Wet") Age-Related Macular Degeneration (NV-AMD)
Brief Title: Safety and Efficacy of ATG003 in Patients With Wet Age-Related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: CoMentis (Industry)
Responsible Party: Carl Grove, CoMentis, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATG003-201
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-10

CONDITIONS: Macular Degeneration
Keywords: AMD; Wet AMD
MeSH Terms: conditions — Macular Degeneration | interventions — Mecamylamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1% mecamylamine (Active Comparator)
  Interventions: Drug: Mecamylamine
- 0.3% mecamylamine (Active Comparator)
  Interventions: Drug: Mecamylamine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mecamylamine
  Arms: 0.3% mecamylamine; 1% mecamylamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase II randomized, double-masked study comparing the safety and efficacy of ATG003 (mecamylamine HCl) 1.0% and 0.3% ophthalmic solutions to placebo in patients with neovascular ("wet") age-related macular degeneration (NV-AMD).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Grove, Study Director — CoMentis
Locations (42):
- Brazil (10):
  - Hospital de Olhos de Araraquara, Araraquara
  - Centro Brasileiro de Ciências Visuais, Belo Horizonte
  - Instituto da Visão, Belo Horizonte
  - Centro Brasileiro de Cirurgia dos Olhos, Goiânia
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro
  - Clínica de Olhos Dr. Suel Abujamra, São Paulo
  - Hospital das Clínicas Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Hospital de Olhos de São Paulo, São Paulo
  - Hospital São Paulo - Setor de Pesquisa Clínica, São Paulo
- Czechia (6):
  - University Hospital Brno, Department of Ophthalmology, Brno
  - Eye Clinic University Hospital, Hradec Králové
  - Ophthalmology Nemocnice Litomysl, Litomyšl
  - University Hospital Olomouc, Department of Ophthalmology, Olomouc
  - Cornea Lexum Praha, Prague
  - Faculty Hospital Kralovske Vinohrady, Dept. of Ophthalmology, Prague
- Mexico (6):
  - Cif Biotec, CP
  - Hospital Conde de Valenciana, CP
  - Fundación Hospital "Nuestra Sra de la Luz" I.A.P., Delegación Cuauhtémoc
  - Asociación Para Evitar la Ceguera, Mexico City
  - Hospital General de México, Mexico City
  - Hospital San José Tec de Monterrey, Monterrey
- Poland (6):
  - Klinika Chorób Oczu, Gdansk
  - Oddział Okulistyczny Okręgowy Szpital Kolejowy, Katowice
  - Klinika Okulistyczna, Lodz
  - Oddział Okulistyki, Samodzielny Publiczny Szpital Kliniczny Nr 1 Przemienienia Pańskiego AM w Poznaniu, Poznan
  - Katedra i Klinika Okulistyki, Samodzielny Publiczny Kliniczny Szpital Okulistyczny, Warsaw
  - Katedra i Klinika Okulistyki, Akademia Medyczna we Wrocławiu, Wroclaw
- Russia (8):
  - Republican Ophthalmologic Hospital of MH of Republic of Tatarstan, Kazan'
  - IRTC "Eye Microsurgery" n. a. S.N. Fyodorov, Moscow
  - Moscow Scientific Research Institute of Eye Diseases, Moscow
  - CJSC "Inter Yuna", Rostov-on-Don
  - City Consultative Diagnostic Centre # 1 (St. Petersburg), Saint Petersburg
  - IRTC "Eye Microsurgery" n. a. S.N. Fyodorov, Saint Petersburg
  - Military Medical Academy n.a. S.M.Kirov of Ministry of Defence, Saint Petersburg
  - St. Petersburg State Medical University n. a. Pavlov, Saint Petersburg
- Ukraine (6):
  - Kyiv City Centre of Eye Vascular and Endocrine Diseases of Organ of Vision, Kyiv
  - Kyiv City Ophthalmologic Hospital "Eye Microsurgery Centre", Kyiv
  - Kyiv City Ophthalmologic Hospital, Kyiv
  - V.P. Filatov Institute of Eye Diseases and Tissue Pathology of AMS of Ukraine, Odesa
  - Zaporizhzhya Center of Vision Rehabilitation, Odesa
  - S.I. Georgiyevsky Crimean State Medical University, Simferopol

REFERENCES:
- See also: Related Info — http://www.comentis.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1% Mecamylamine | 0.3% Mecamylamine | Placebo
Started | 115 | 114 | 114
Completed | 57 | 58 | 59
Not Completed | 58 | 56 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Mecamylamine | 0.3% Mecamylamine | Placebo | Total
Number analyzed (Participants) | 115 | 114 | 114 | 343
Age Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8) | 72.6 (8.7) | 71.3 (7.7) | 72.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 71 | 77 | 213
  Male | 50 | 43 | 37 | 130
Region of Enrollment [Number; unit: participants]
  Czech Republic | 11 | 15 | 12 | 38
  Mexico | 7 | 7 | 6 | 20
  Brazil | 15 | 13 | 16 | 44
  Poland | 19 | 21 | 17 | 57
  Ukraine | 34 | 32 | 35 | 101
  Russian Federation | 26 | 26 | 28 | 80
  United States | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Losing Fewer Than 15 ETDRS Letters of Visual Acuity at 48 Weeks Compared to Baseline.
Time Frame: Baseline to Week 48
Population: A modified MITT population was used, which was prospectively defined as all randomized patients who received at least one dose of study drug and had at least one post-baseline efficacy (visual acuity) assessment.
Measure: Number; unit: Percent of subjects
Arm/Group | 1% Mecamylamine | 0.3% Mecamylamine | Placebo
Number analyzed (Participants) | 113 | 112 | 113
Percent of subjects | 88 | 86 | 92
Statistical Analysis 1: Comparison: 1% Mecamylamine vs 0.3% Mecamylamine vs Placebo; Test type: Superiority or Other; p > 0.05, ANCOVA

ADVERSE EVENTS:
Arm/Group | 1% Mecamylamine | 0.3% Mecamylamine | Placebo
Serious Adverse Events (participants affected / at risk) | 8/115 | 8/115 | 7/114
Other Adverse Events (participants affected / at risk) | 68/115 | 57/114 | 57/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% Mecamylamine (N=115) | 0.3% Mecamylamine (N=115) | Placebo (N=114)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal ucler (General disorders) | 0 (0) | 0 (0) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1% Mecamylamine (N=115) | 0.3% Mecamylamine (N=114) | Placebo (N=114)
Cardiac disorders (Cardiac disorders) | 4 (4) | 8 (8) | 4 (4)
Visual acuity reduced (Eye disorders) | 38 (38) | 31 (31) | 38 (38)
Retinal haemorrhage (Eye disorders) | 17 (17) | 11 (11) | 16 (16)
Cataract (Eye disorders) | 7 (7) | 0 (0) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 9 (9) | 5 (5) | 8 (8)
Infections and Infestiations (Infections and infestations) | 19 (19) | 16 (16) | 12 (12)
Investigations (Investigations) | 4 (4) | 6 (6) | 7 (7)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 4 (4)
Nervous system disorders (Nervous system disorders) | 15 (15) | 2 (2) | 9 (9)
Headache (Nervous system disorders) | 6 (6) | 2 (2) | 4 (4)
Vascular disorders (Vascular disorders) | 6 (6) | 3 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less